CLINICAL TRIAL: NCT01004523
Title: Diagnostic and Prognostic Markers in Low-Grade Gliomas
Brief Title: Study of Tissue and Blood Samples From Patients With Low-Grade Glioma
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCCTG-94-72-53; NCCTG-947253; CDR0000406626 (Registry Identifier: PDQ (Physician Data Query)); NCI-2009-00689 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood low-grade cerebellar astrocytoma; childhood low-grade cerebral astrocytoma; childhood mixed glioma; adult mixed glioma; adult diffuse astrocytoma; childhood oligodendroglioma; adult oligodendroglioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioma; Astrocytoma; Oligodendroglioma | interventions — In Situ Hybridization, Fluorescence; Polymerase Chain Reaction; Flow Cytometry; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissue and blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single group: Previously preserved paraffin-embedded tissue blocks are obtained and used for biomarker studies. Blood samples obtained during treatment are also obtained. Loss of heterozygosity of specific chromosomal regions are performed using PCR analysis of microsatellite repeats (41,118-120) on DNA extracted from the paraffin-embedded archival specimens. FISH and flow cytometry may also be used to assess chromosomal loss of deletion. Immunohistochemistry is also performed.
  Interventions: Genetic: fluorescence in situ hybridization; Genetic: loss of heterozygosity analysis; Genetic: polymerase chain reaction; Other: flow cytometry; Other: immunohistochemistry staining method

INTERVENTIONS:
Genetic: fluorescence in situ hybridization
Genetic: loss of heterozygosity analysis
Genetic: polymerase chain reaction
Other: flow cytometry
Other: immunohistochemistry staining method

SUMMARY:
RATIONALE: Studying samples of tumor tissue and blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is looking at tissue and blood samples from patients with low-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the diagnostic and prognostic relevance of alterations of specific chromosomes and chromosomal regions including 7, 9p, 10p, 10q, 13q, 17p, 17q, 19q, 22q, X, and Y, using PCR analysis of microsatellite repeats and FISH.
* Evaluate the diagnostic and prognostic relevance of DNA ploidy by flow cytometric analysis; compare with ploidy determination by FISH.
* Assess the diagnostic and prognostic relevance of various markers of cellular proliferation and cellular function including flow cytometric determination of %S-phase, %G2M, and immunohistochemical evaluation of PCNA, Ki-67, and p53.

ELIGIBILITY:
1. Paraffin-embedded tumor tissue blocks of patients enrolled in NCCTG 86-72-51 or 93-72-02 and who had the diagnosis of low-grade glioma.
2. Patients who have the diagnosis of low-grade glioma with an available paraffin- embedded tumor tissue block enrolled in prospective NCCTG and Mayo studies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with low grade glioma.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 1995-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Alterations in chromosomes 7, 9p, 10, 17, 19q, X, or Y as determined by FISH | baseline
Loss of chromosomal materials in chromosomes 9p, 10, 13, 17, or 22 by PCR analysis | baseline
Levels of PCNA, Ki-67 (MIB-1), or mutated p53 by immunostaining with monoclonal antibodies | baseline
DNA ploidy by FISH and flow cytometry | baseline
Percentage of cells in S-phase or G2M-phase as measured by flow cytometry | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jan Buckner, MD, Study Chair — Mayo Clinic
Locations (38):
- United States (38):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Essentia Health - Duluth Clinic, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia